CLINICAL TRIAL: NCT02303522
Title: A Retrospective Pooled Analysis of Complete Remission Among Pediatric Patients With Relapsed or Refractory B-cell Precursor Acute Lymphoblastic Leukemia (ALL)
Brief Title: Historical Data Analysis of Complete Remission in Children With R/R Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120299
Record Dates: First submitted 2014-11-06; First posted 2014-12-01 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: B-cell Precursor Acute Lymphoblastic Leukemia (ALL)
Keywords: ALL, pediatric, leukemia, childhood, lymphoblastic, lymphoma, acute, Precursor Cell
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All subjects: All subjects will be included in a unique cohort
  Interventions: Other: Other: not applicable - observational study

INTERVENTIONS:
Other: Other: not applicable - observational study — No intervention exists as this is a retrospective observational study

SUMMARY:
An historical data comparator study for children with relapsed/refactory acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
A retrospective observational study reviewing historical complete remission for pediatric patients who had either relapsed or refractory B-precursor acute lymphoblastic leukemia (ALL)

ELIGIBILITY:
Inclusion criteria:

* Pediatric (age less than 18 years) patients with relapsed or refractory B-cell precursor ALL, specifically those with
* 2nd or later relapse after chemotherapy (with no prior transplantation),
* Relapse after HSCT, or
* Refractory disease
* Had treatment for relapsed or refractory disease between 2005-2012
* Has data available on ALL treatment, including number of salvage treatments, response status after therapies, and HSCT

Exclusion criteria:

* No CNS involvement at relapse
* No previous treatment with blinatumomab

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with relapsed or refractory B-cell precursor acute lymphoblastic leukemia (ALL)
Sampling Method: Non-Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2014-12-09 (Actual); Primary Completion 2015-01-22 (Actual); Study Completion 2015-01-22 (Actual)

PRIMARY OUTCOMES:
Hematological Complete Remission (CR) | Approx. 1 year
  To estimate hematological Complete Remission (CR) in pediatric patients with relapsed or refractory B-cell precursor Acute Lymphoblastic Leukemia (ALL)

SECONDARY OUTCOMES:
Overall survival | Approx. 1 year
  OS following salvage therapy: defined as time to death.
Molecular CR | Approx. 1 year
  Defined as MRD <10-4 measured either by PCR or flow cytometry.
Relapse Free Survival (RFS) | Approx. 1 year
  Defined as time to relapse or death.
Time to hematological CR | Approx. 1 year
  Defined as time to unequivocal detection of >5% leukemia cells in bone marrow as measured by cytological, microscopic assessment, presence of circulating leukemia blasts, or extramedullary leukemia
Receipt of HSCT after salvage treatment | Approx. 1 year
  Defined as the receipt of HSCT after chemotherapy or a previously failed HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- Research Site, Vienna, Austria
- Research Site, Berlin, Germany
- Research Site, Roma, Italy

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com